CLINICAL TRIAL: NCT07396922
Title: A Randomized, Controlled Study to Evaluate the Efficacy and Safety of the SSMD in Neuromotor Rehabilitation
Brief Title: Assessment of Safety and Effectiveness of Spatial StimelMD (SSMD) in Subjects With Upper Limb Neuromotor Impairments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motion Informatics LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-SSMD-02
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stroke; TBI; Spinal Cord Injury; Peripheral Nerve Damage
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Neuritis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) into two parallel groups to receive either SSMD plus conventional therapy or FES plus conventional therapy
Masking Description: This is an open-label study. No masking/blinding is implemented due to the nature of the device interventions and treatment delivery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- SSMD + Conventional Therapy (Experimental): Participants receive SSMD sessions in addition to conventional therapy for 18 sessions (30 minutes each), delivered 6 sessions per week over 3 weeks.
  Interventions: Device: SSMD
- FES + Conventional Therapy (Active Comparator): Participants receive functional electrical stimulation (FES) sessions in addition to conventional therapy for 18 sessions (30 minutes each), delivered 6 sessions per week over 3 weeks.
  Interventions: Device: Functional Electrical Stimulation (FES)

INTERVENTIONS:
Device: SSMD — SSMD device-based therapy delivered in addition to conventional therapy. Participants receive 18 sessions, 30 minutes each, administered 6 sessions per week over 3 weeks.
  Arms: SSMD + Conventional Therapy
Device: Functional Electrical Stimulation (FES) — Functional electrical stimulation (FES) delivered in addition to conventional therapy. Participants receive 18 sessions, 30 minutes each, administered 6 sessions per week over 3 weeks.
  Arms: FES + Conventional Therapy

SUMMARY:
This study will evaluate the safety and performance of the Spatial StimeMD (SSMD) medical device in people with multiple sclerosis (MS). The SSMD device is intended to support patients through a non-invasive stimulation program. The study will assess changes in MS-related symptoms and physical function using clinical assessments and patient-reported outcomes.

DETAILED DESCRIPTION:
This is a clinical investigation of the Spatial StimeMD (SSMD) medical device in participants diagnosed with multiple sclerosis (MS). The purpose of the study is to evaluate the safety and performance of the device in a controlled clinical setting. Participants will be followed according to the study schedule and will undergo assessments of MS symptoms, physical function, and other relevant clinical outcomes. Safety will be assessed through monitoring of adverse events and other safety parameters throughout the study. Study data will be collected and reviewed according to the protocol, including verification against source documentation as required.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 18-80 years.
2. Clinically confirmed diagnosis of stroke, TBI, spinal cord injury, or peripheral nerve injury within the past 24 months.
3. Presence of moderate to severe neuromotor impairment in at least one limb, as evidenced by medical evaluation and a score <35 on the Fugl-Meyer Upper Extremity motor subscale (FMA-UE).
4. Capacity and willingness to provide informed consent, indicating understanding of the study purpose, procedures, and potential risks and benefits.
5. Subject is able to adhere to the study schedule and cognitively capable to perform the treatment.
6. Stable medical condition without ongoing acute complications that could interfere with participation.

Exclusion Criteria:

1. Presence of contraindications to electrical stimulation (ES), including implanted electronic medical devices (e.g., Cardiac demand pacemakers, Implantable pacemakers, Implantable cardioverter defibrillators, Implantable neurostimulators, Body-worn devices such as insulin pumps) or conditions that may be exacerbated by electrical stimulation (e.g., uncontrolled epilepsy).
2. Individuals with medical conditions, which are prone to seizures or motion sensitivity, at the investigator's discretion.
3. Individuals with light sensitivity, as the AR component may involve visual stimuli that could cause discomfort or adverse reactions in these patients.
4. Individuals with acute physical conditions or injuries that could interfere with the proper placement of the electrodes or safe use of the device.
5. Presence of spinal shock or unresolved acute spinal cord dysfunction, characterized by complete loss of reflexes, flaccid paralysis, or autonomic instability.
6. Current participation in other clinical trials that could confound the study results.
7. Severe cognitive impairment that precludes the ability to provide informed consent or reliably adhere to the study protocol, as determined by cognitive screening and clinical judgment.
8. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Upper Extremity (FMA-UE) motor score | Baseline to post-treatment (end of treatment, 3 weeks)
  Change from baseline in Fugl-Meyer Assessment Upper Extremity (Motor Function Subscale) The Fugl-Meyer Assessment Upper Extremity motor score is a clinician-rated measure of upper limb motor impairment following neurological injury. Scores range from 0 to 66, with higher scores representing less impairment and better motor function.
  Time Frame: Baseline to post-treatment (3 weeks).

SECONDARY OUTCOMES:
change in Movement range and movement quality (SSMD assessment mode) | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in movement range and movement quality as assessed using the SSMD system assessment mode.
Change in Functional Independence Measure (FIM) score | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in activities of daily living as measured by the Functional Independence Measure (FIM) total score (range 18-126, higher scores indicate greater independence and better functional outcome).
  Time Frame: Baseline to end of treatment (Week 3).
Change in EMG signal strength (threshold) | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in electromyography (EMG) signal strength (threshold) during device-assisted assessment.

OTHER OUTCOMES:
Change in Modified Ashworth Scale (MAS) | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in spasticity as measured by the Modified Ashworth Scale (range 0-4; higher scores indicate greater spasticity and worse outcome).
  Time Frame: Baseline to end of treatment (Week 3).
Change in Stroke Impact Scale (SIS) score | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in Stroke Impact Scale (SIS) score (range 0-100; higher scores indicate better function and less stroke impact).
  Time Frame: Baseline to end of treatment (Week 3).
Change in NIH Stroke Scale (NIHSS) score | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in National Institutes of Health Stroke Scale (NIHSS) score (range 0-42; higher scores indicate more severe neurologic deficit and worse outcome).
  Time Frame: Baseline to end of treatment (Week 3).
Change in Active Range of Motion (AROM) measured by goniometer | Baseline to post-treatment (end of treatment, Week 3)
  Change from baseline to post-treatment in active range of motion (AROM) (0-70 degrees), measured by goniometer.
System Usability Scale (SUS) score | Post-treatment (end of treatment, Week 3)
  System usability assessed by the System Usability Scale (SUS) (range 0-100; higher scores indicate better usability).
  Time Frame: Post-treatment (Week 3).
Adverse events (AEs) | Baseline through end of follow-up (up to 6 weeks)
  Frequency and severity of all adverse events (AEs), related or unrelated to study treatment.
Observer usability questionnaire score | Post-treatment (end of treatment, Week 3)
  Observer-reported usability will be assessed using a custom Observer Usability Questionnaire evaluating effectiveness and efficiency of device use (e.g., task accuracy, ease of navigation, and assistance required). Questionnaire items are rated on a 5-point scale (1 = poorest performance/usability, 5 = best performance/usability). An overall usability score will be calculated as the mean of the rated items, with higher scores indicating better usability and task performance.
  Time Frame: Post-treatment (end of treatment, Week 3).

CONTACTS AND LOCATIONS:
Locations (1):
- Polsko-Amerykańskie Kliniki Serca SA, Uzdrowisko Ustroń, Ustroń, Poland

IPD SHARING:
Plan to Share IPD: Undecided